CLINICAL TRIAL: NCT06375603
Title: Nerve and Plane Block Data Collection Study for the Development of Artificial Intelligence-assisted Software
Status: Completed | Type: Observational
Sponsor: Smart Alfa Teknoloji San. ve Tic. A.S. (Industry)
Collaborators: Ankara University (Other)
Responsible Party: Sponsor
Other Study IDs: SMARTALPHA-NERVEBLOX-1001
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Ultrasound Imaging of Anatomical Structures; Nerve Block
Keywords: Ultrasound Imaging; Artificial Intelligence; Nerve Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ultrasound scans — Clinical experts will conduct non-invasive ultrasound scans from the specified nerve or plane block views and record the acquired data.

SUMMARY:
The primary objective of this observational study is to acquire ultrasound images (raw data) from nerve and plane block regions to develop artificial intelligence-guided nerve block software (Nerveblox). The study aims to acquire raw ultrasound video from 200 volunteers' planned nerve and plane block regions. These participants will undergo ultrasound scans administered by expert clinicians proficient in these techniques in their clinical practice. The data collection devices utilized in this study are FDA-cleared general-purpose ultrasound devices.

DETAILED DESCRIPTION:
Ultrasound-guided nerve and plane blocks have facilitated regional anesthesia by providing clinicians with real-time imaging capabilities for precise needle placement and application of local anesthetics. These techniques involve the use of ultrasound technology to visualize nerves and surrounding anatomical structures, allowing for accurate identification and targeting of specific nerve pathways. Additionally, the integration of artificial intelligence (AI) into ultrasound-guided nerve blocks offers further enhancements to this practice. AI algorithms can assist clinicians in image interpretation, needle localization, and decision-making, streamlining procedural workflows and reducing the risk of complications. The sponsor, Smart Alfa Teknoloji San. Ve Tic. A.Ş., located in Ankara, Turkey, aims to collect data from planned regions of volunteers to develop artificial intelligence-supported nerve block software (Nerveblox). The gathered data will be utilized for training, validation, and test processes of the AI algorithm.

The study methodology encompasses the following components:

* A cohort of 200 volunteers, evenly distributed by gender (100 male, 100 female), will have their demographic data (BMI, gender, age) documented.
* Each scan from one volunteer is expected to take 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Male at least 18 years of age
* Female at least 18 years of age
* Health volunteers
* Able to confirm and sign the Informed Consent Form before enrolment the study

Exclusion Criteria:

* Male below 18 years of age
* Female below 18 years of age
* Unwilling to participate or unable to sign an informed consent form
* Inability to lie flat
* Anatomical deformity in the area to be scanned for nerve and plane blocks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200 healthy volunteers will participate in the data collection study. Their weight, height, age, and gender information will be documented.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Assessment of image quality | 6 months
  Collected images will be used for labeling anatomical landmarks for development of Nerveblox.

CONTACTS AND LOCATIONS:
Overall Officials: Süheyla Karadağ Erkoç, Assoc. Prof., Principal Investigator — Ankara University
Locations (1):
- Ankara University School of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No